CLINICAL TRIAL: NCT02441374
Title: Efficacy of Modified FUT Protocols With 12 and 24 Hours of Upper Limb Immobilization in Relation to CR Arm Protocol.
Brief Title: Efficacy of Modified FUT Protocols in Relation to CR Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Tamyris Padovani dos Santos, João Eduardo de Araujo, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TPSantos
Record Dates: First submitted 2015-04-09; First posted 2015-05-12 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: Stroke; Hemiparesis; Upper limb
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Forced Use Therapy (Experimental): Constriction (through the tubular mesh) of non paretic upper limb for a period of 12 and 24 hours, 5 days per week for 4 weeks.
  Interventions: Device: Tubular mesh.
- Classical Kinesiotherapy (Active Comparator): Rehabilitation of classical kinesiotherapy,at least 2 times a week for 4 weeks.
  Interventions: Other: Classical kinesiotherapy.

INTERVENTIONS:
Device: Tubular mesh. — Rehabilitation in upper limb during and after applying of FUT (through the tubular mesh) post stroke.
  Arms: Forced Use Therapy
Other: Classical kinesiotherapy. — Applying classical kinesiotherapy in upper limb post stroke.
  Arms: Classical Kinesiotherapy

SUMMARY:
There are some treatments after Stroke. Among these, use forced therapy (FUT), which is based on overcoming learned disuse by reintroduction of the paretic upper limb in the performance of daily activities. There are different protocols FUT to the daily time constraint, the number of days and even the type of constriction. Researchers have developed a protocol using four weeks constriction, daily constriction 24 hours and with the free end of the weekends. Because it is a restrictive therapy, which requires the use of one of the arms and on the other hand, this mode of treatment is open to criticism, however, despite the efficacy of the protocol, patients do not have good adhesion to the protocol for the constriction severe over time. The objective of this work is to verify the safety of the developed protocol and analyze the feasibility of reducing the daily time of constriction 12 hours, with a new protocol movement constriction, easier to perform and more patient acceptance. Participate in this study 82 individuals hemiparetic post Stroke, which will be recruited to Neurovascular Diseases Clinic and will be registered at the Rehabilitation Center of Integrated State Hospital. Participants will be randomly divided into three groups: the FUT24 (non-paretic upper limb constriction 24 hours a day, five days a week for 4 weeks), the FUT 12 (non-paretic upper limb constriction for 12 hours a day, five days a week for 4 weeks) and CK (Classic Kinesiotherapy, at least 2 times a week for 4 weeks). Will be held weekly and after the end of the monthly monitoring reviews protocols. For the rating scales are use: National Institute of Health Stroke Scale, the Ashworth Scale, the Wolf Motor Function Test, the Motor Activity Log, Fugl-Meyer Assesment, dynamometry handgrip and surface electromyography (flexor and extensor muscles wrist). The researchers hope that this protocol does not bring damage to the upper limb in constriction and it is established a new protocol FUT easier to perform and more acceptable to patients, allowing the use of this technique by health professionals.

DETAILED DESCRIPTION:
The constriction of the non-paretic upper limb will be conducted through a tubular mesh with UL positioned in adduction and shoulder internal rotation and elbow flexion greater than 90º in FUT 24 and FUT 12 groups. Daily, the mesh is withdrawn by the investigators made hygienic, and the new constraint is accomplished using a new tubular mesh.The Classic Kinesiotherapy Group,which will receive as a treatment only kinesiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Good cognition,
2. Absence of joint blocks,
3. Good range of motion in upper limb with at least 20º of active extension of the wrist and 10º in the metacarpal phalangeal,
4. Joint and walking capacity without assistance.

Exclusion Criteria:

1. Heart arrhythmia,
2. Hypertension,
3. Severe cardiovascular and respiratory problems,
4. Inability to attend the sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of RMS activity through surface electromyography. | 4 months
  Evaluations shall be performed weekly during the treatment period and 1 monthly assessment for 3 months after the protocol without therapeutic intervention.

SECONDARY OUTCOMES:
Evaluate the strength handgrip (Kgf) of hemiparetic patients submitted to FUT post stroke. | 4 months
  Evaluations shall be performed weekly during the treatment period and 1 monthly assessment for 3 months after the protocol without therapeutic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tamyris Padovani dos Santos, Principal Investigator — University of Sao Paulo
Locations (1):
- Tamyris Padovani dos Santos, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmed S, Mayo NE, Higgins J, Salbach NM, Finch L, Wood-Dauphinee SL. The Stroke Rehabilitation Assessment of Movement (STREAM): a comparison with other measures used to evaluate effects of stroke and rehabilitation. Phys Ther. 2003 Jul;83(7):617-30. PMID 12837123
- [Result] Brown MM. Brain attack: a new approach to stroke. Clin Med (Lond). 2002 Jan-Feb;2(1):60-5. doi: 10.7861/clinmedicine.2-1-60. PMID 11871641
- [Result] Brott T, Adams HP Jr, Olinger CP, Marler JR, Barsan WG, Biller J, Spilker J, Holleran R, Eberle R, Hertzberg V, et al. Measurements of acute cerebral infarction: a clinical examination scale. Stroke. 1989 Jul;20(7):864-70. doi: 10.1161/01.str.20.7.864. PMID 2749846
- [Result] Cincura C, Pontes-Neto OM, Neville IS, Mendes HF, Menezes DF, Mariano DC, Pereira IF, Teixeira LA, Jesus PA, de Queiroz DC, Pereira DF, Pinto E, Leite JP, Lopes AA, Oliveira-Filho J. Validation of the National Institutes of Health Stroke Scale, modified Rankin Scale and Barthel Index in Brazil: the role of cultural adaptation and structured interviewing. Cerebrovasc Dis. 2009;27(2):119-22. doi: 10.1159/000177918. Epub 2008 Nov 28. PMID 19039215
- [Result] Charles J, Gordon AM. A critical review of constraint-induced movement therapy and forced use in children with hemiplegia. Neural Plast. 2005;12(2-3):245-61; discussion 263-72. doi: 10.1155/NP.2005.245. PMID 16097492
- [Result] Cirstea MC, Levin MF. Improvement of arm movement patterns and endpoint control depends on type of feedback during practice in stroke survivors. Neurorehabil Neural Repair. 2007 Sep-Oct;21(5):398-411. doi: 10.1177/1545968306298414. Epub 2007 Mar 16. PMID 17369514
- [Result] De Marchis GM, Foderaro G, Jemora J, Zanchi F, Altobianchi A, Biglia E, Conti FM, Monotti R, Mombelli G. Mild cognitive impairment in medical inpatients: the Mini-Mental State Examination is a promising screening tool. Dement Geriatr Cogn Disord. 2010;29(3):259-64. doi: 10.1159/000288772. Epub 2010 Apr 6. PMID 20375507
- [Result] De D, Wynn E. Preventing muscular contractures through routine stroke patient care. Br J Nurs. 2014 Jul 24-Aug 13;23(14):781-6. doi: 10.12968/bjon.2014.23.14.781. PMID 25062313
- [Result] Feigin VL, Barker-Collo S, Krishnamurthi R, Theadom A, Starkey N. Epidemiology of ischaemic stroke and traumatic brain injury. Best Pract Res Clin Anaesthesiol. 2010 Dec;24(4):485-94. doi: 10.1016/j.bpa.2010.10.006. Epub 2010 Nov 29. PMID 21619861
- [Result] Fuzaro AC, Guerreiro CT, Galetti FC, Juca RB, Araujo JE. Modified constraint-induced movement therapy and modified forced-use therapy for stroke patients are both effective to promote balance and gait improvements. Rev Bras Fisioter. 2012 Apr;16(2):157-65. doi: 10.1590/s1413-35552012005000010. Epub 2012 Mar 1. PMID 22378476
- [Result] Green J, Forster A, Young J. Reliability of gait speed measured by a timed walking test in patients one year after stroke. Clin Rehabil. 2002 May;16(3):306-14. doi: 10.1191/0269215502cr495oa. PMID 12017517
- [Result] Hagg S, Thorn LM, Forsblom CM, Gordin D, Saraheimo M, Tolonen N, Waden J, Liebkind R, Putaala J, Tatlisumak T, Groop PH; FinnDiane Study Group. Different risk factor profiles for ischemic and hemorrhagic stroke in type 1 diabetes mellitus. Stroke. 2014 Sep;45(9):2558-62. doi: 10.1161/STROKEAHA.114.005724. Epub 2014 Jul 24. PMID 25061078
- [Result] Lavados PM, Hennis AJ, Fernandes JG, Medina MT, Legetic B, Hoppe A, Sacks C, Jadue L, Salinas R. Stroke epidemiology, prevention, and management strategies at a regional level: Latin America and the Caribbean. Lancet Neurol. 2007 Apr;6(4):362-72. doi: 10.1016/S1474-4422(07)70003-0. PMID 17362840
- [Result] Liepert J, Uhde I, Graf S, Leidner O, Weiller C. Motor cortex plasticity during forced-use therapy in stroke patients: a preliminary study. J Neurol. 2001 Apr;248(4):315-21. doi: 10.1007/s004150170207. PMID 11374097
- [Result] Michaelsen SM, Rocha AS, Knabben RJ, Rodrigues LP, Fernandes CG. Translation, adaptation and inter-rater reliability of the administration manual for the Fugl-Meyer assessment. Rev Bras Fisioter. 2011 Jan-Feb;15(1):80-8. PMID 21519719
- [Result] Mark VW, Taub E, Morris DM. Neuroplasticity and constraint-induced movement therapy. Eura Medicophys. 2006 Sep;42(3):269-84. PMID 17039225
- [Result] Taub E, Uswatte G, King DK, Morris D, Crago JE, Chatterjee A. A placebo-controlled trial of constraint-induced movement therapy for upper extremity after stroke. Stroke. 2006 Apr;37(4):1045-9. doi: 10.1161/01.STR.0000206463.66461.97. Epub 2006 Mar 2. PMID 16514097
- [Result] Scherbakov N, von Haehling S, Anker SD, Dirnagl U, Doehner W. Stroke induced Sarcopenia: muscle wasting and disability after stroke. Int J Cardiol. 2013 Dec 10;170(2):89-94. doi: 10.1016/j.ijcard.2013.10.031. Epub 2013 Oct 14. PMID 24231058
- [Result] Taub E, Uswatte G. Constraint-induced movement therapy: bridging from the primate laboratory to the stroke rehabilitation laboratory. J Rehabil Med. 2003 May;(41 Suppl):34-40. doi: 10.1080/16501960310010124. PMID 12817655
- [Result] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415